CLINICAL TRIAL: NCT00013377
Title: Predictors of Driving Performance and Successful Mobility - Rehabilitation in Patients With Medical Eye Condition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: C1982R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Low Vision
Keywords: Low vision, Driving rehabilitation
MeSH Terms: conditions — Vision, Low

INTERVENTIONS:
Procedure: Low vision

SUMMARY:
There are two diseases in particular that may have serious consequences for driving and mobility due to their potentially severe impact on visual function: glaucoma and diabetic neuropathy. In this project we will develop predictive models of driving for these patients and will train them to use low-vision aids to improve driving mobility. We will determine how best to train patients with hemianopic field loss due to cerebral vascular accidents and identify predictors of long-term success in the use of low-vision aids.

DETAILED DESCRIPTION:
There are two diseases in particular that may have serious consequences for driving and mobility due to their potentially severe impact on visual function: glaucoma and diabetic neuropathy. Both these diseases can potentially result in significant peripheral visual field loss, sometimes coupled with decreased visual acuity. We have previously demonstrated that each of these visual losses alone can have significant impact on driving and mobility performance. In this project we will develop predictive models of driving for these patients and apply our extensive expertise in training patients to use low-vision aids to improve driving mobility. A second question that will be addressed is how to best train scanning patients with hemianopic field loss due to cerebral vascular accidents. We propose to configure the prisms in a bioptic form similar to previously used for amorphic lenses in RP and for bioptic telescopes for patients in macular disease. The third problem that will be addressed is the identification of predictors of long-term success in the use of low-vision aids.

ELIGIBILITY:
Eye impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1999-04; Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph. D., Asst. Director — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Nancy Rocheleau, Program Analyst — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC (West Side), Chicago, Illinois, United States